CLINICAL TRIAL: NCT02153840
Title: A Double-blind, Randomized, Placebo-controlled Trial of PSORI-CM01（YXBCM01） Granule for Stable Plaque Psoriasis
Brief Title: Clinical Trial of PSORI-CM01（YXBCM01） Granule to Treat Stable Plaque Psoriasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Paitents were unwilling to be randomly assigned to a placebo group.
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chuanjian Lu, Doctor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201105
Record Dates: First submitted 2014-05-24; First posted 2014-06-03 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Plaque Psoriasis
Keywords: Stable Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PSORI-CM01（YXBCM01）granule (Experimental): PSORI-CM01（YXBCM01）granule 1.1g os once a day for 12weeks.
  Interventions: Drug: PSORI-CM01（YXBCM01） granule
- PSORI-CM01（YXBCM01）granule low dose group (Experimental): PSORI-CM01（YXBCM01） granule 5.5g os once a day for 12weeks.
  Interventions: Drug: PSORI-CM01（YXBCM01） granule; Drug: placebo
- placebo (Placebo Comparator): Placebo granule 1.1g os once a day for 12weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PSORI-CM01（YXBCM01） granule
  Other Names: Chinese Hebal Medicine
  Arms: PSORI-CM01（YXBCM01）granule; PSORI-CM01（YXBCM01）granule low dose group
Drug: placebo
  Arms: PSORI-CM01（YXBCM01）granule low dose group; placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Chinese herbal PSORI-CM01（YXBCM01） granule for stable plaque psoriasis, with blood stasis syndrome of Chinese Medicine.

DETAILED DESCRIPTION:
Psoriasis is an immune-abnormal, chronic, proliferative skin disease characterized by scaly, erythematous patches and papules. An epidemiological survey found Chinese prevalence showed an upward trend in recent years. The disease has great influence on patients' appearance,health and quality of life. Some Chinese Herbal Medicine (CHM) therapies have shown long lasting therapeutic effect on controlling psoriasis vulgaris and with minimal side effects.CHM can alleviate the symptoms effectively,and reduce the recurrence rate of diseases. PSORI-CM01（YXBCM01）granule is one kind of CHM which is observed effective and safe to treat stable stable plaque psoriasis with blood stasis syndrome in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Stable plaque psoriasis, duration > 1 year.
2. Patients with Chinese medicine blood stasis syndrome. (2)18 to 65 years old, male or female patient.
3. Mild psoriasis:3<PASI≤10, and BSA≤10%.
4. Informed consent.

Exclusion Criteria:

1. Guttate psoriasis, inverse psoriasis or exclusively involves the face;
2. Acute progression of psoriasis, and erythroderma tendency.Not blood stasis syndrome.Not stable psoriasis.
3. Pregnant, lactating, or which one plan to become pregnant in a year;
4. SAS（Self-rating Anxiety Scale）> 50 or SDS（Self-rating Depression Scale）> 53, or with other psychiatric disorders;
5. With history of cardiovascular, respiratory, digestive, urinary, and hematologic disease, which can't controlled through common treatment. Either with cancer, infection, electrolyte imbalance, acid-base disturbance and calcium metabolic disorder.
6. Allergic to any medicine or ingredients used in this study.
7. Participating other clinical trials or participated within 1 month.
8. Topical treatments (i.e. corticosteroids, Retinoic acid) within 2 weeks; systemic therapy or phototherapy (UVB and PUVA) within 4 weeks; biological therapy within 12 weeks.
9. Patients need systemic treatment prescribed by doctors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
PASI-50 | 12 weeks (plus or minus 3 days) after treatment
  The number of patients who achieve at least 50% improvement in PASI score from baseline.

SECONDARY OUTCOMES:
PASI(Psoriasis Area and Severity Index) | 12 weeks (plus or minus 3 days) after treatment
  The improvement in PASI score from baseline.
PASI-75 | 12 weeks (plus or minus 3 days) after treatment
  The number of patients who achieve at least 75% improvement in PASI score from baseline.
Pruritus Scores on the Visual Analogue Scale | 12 weeks (plus or minus 3 days) after treatment
BSA（Body Surface Area） | 12 weeks (plus or minus 3 days) after treatment
  the Body Surface Area
DLQI（Dermatology Life Quality Index） | 12 weeks (plus or minus 3 days) after treatment
  the Dermatology Quality Life Index
Relapse rate in treatment period / follow-up period | During the treatment period of 12 weeks / follow-up period of 12 weeks after treatment period
  Relapse can be defined only for patients who achieve PASI50，and occurs when the improvement in the PASI score falls below 50% from the baseline PASI score.
Time interval for patients the first time to achieve PASI-50 from baseline | During the treatment period of 12 weeks
Relapse time interval | During the treatment period of 12 weeks / follow-up period of 12 weeks after treatment period
  Relapse time interval refers to the time when patients who achieve PASI-50 for the first time until first relapse occurs.
Rebound rate | During the treatment period of 12 weeks / follow-up period of 12 weeks after treatment period
  Rebound can be defined only for patients who achieve PASI50，and occurs when the improvement in the PASI score increase up to 25% from the baseline PASI score.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjian Lu, Doctor, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - Chronic Disease Prevention and Control Station of Panyu District in Guangzhou, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong